CLINICAL TRIAL: NCT05751447
Title: Studie Av Cellulära Uttryck I Lymfkörtlar, Lungsköljvätska Och Blod Vid Sarkoidos.
Brief Title: Sarcoidosis and Immune Cells in Lung, Lymph Nodes and Blood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K2019-6557
Record Dates: First submitted 2023-02-06; First posted 2023-03-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immune cells (Experimental): Lymph node puncture and/ or bronchoscopy.
  Interventions: Diagnostic Test: Lymph node puncture, bronchoscopy

INTERVENTIONS:
Diagnostic Test: Lymph node puncture, bronchoscopy — Included patients will undergo an extra lympn node punction through oesophagus and/ or an extra bronchoscopy.

SUMMARY:
Background:

Sarcoidosis is an inflammatory disease, most commonly affecting the lungs and intrathoracic lymph nodes but can affect virtually any organ, sometimes manifesting as life threatening cardiac arrythmias. Some patients resolve spontaneously, whereas others get a chronic disease leading to for instance impaired lung function and cardiac failure. The most severe cases might need a transplantation.

In the lungs, activated T cells are accumulated leading to release of cytokines, especially TNF-alpha is regarded as crucial for disease progression. Some segments of the T cell receptor and specific genes (HLA types) are connected to a resolving disease. More detailed knowledge about mechanisms why some experience a chronic disease course and others resolve spontaneously without treatment is to a large extent lacking. There is no cure, and despite treatment with immunosuppressants (often corticosteroids and cytotoxic agents), many patients experience a deteriorating disease.

Aim:

1. Find biomarkers to be able to early predict which patients will develop a more severe/ chronic disease course and thereby enabeling early intervention before irreversible damage.
2. Predict which treatment is best for a specific patient, i.e. individualize treatment.
3. Find targets for new potential therapies.

Methods:

The majority of data is collected at investigations normally performed during diagnostic work-up for sarcoidosis. Most patients undergo a bronchoscopy with bronchoalveolar lavage (BAL) and some also lymph node punction through oesophagus with the help of ultrasound. The BAL fluid that remains after clinical analysis is used for research purpose. For patients undergoing lymph node punction, one extra punction is performed for research purpose. Extra blood samples are taken from all patients.

The samples will mostly be used for studying T cells with immunohistochemistry, flow cytometry including activity markers, subtypes and receptors, but also cytokines and other cells (for instance B cells, NK and NKT cells). The patients are followed longitudinally, minimum 2 years. Some patients will undergo a second bronchoscopy 6-12 months after the first. Results from the immunological investigations will be correlated to disease course, genetics and result of treatment.

Significance :

By comparing the inflammation in several compartments (lung, lymph node , blood) at a molecular level with clinical disease course, genotype, and treatment response we hope to find biomarkers that can predict disease course and response to therapy. Thereby, we hope to be able to tailor therapy for each individual patient. By studying several compartments, the results may also help to improve understanding of how a systemic inflammation is distributed within the body, and thus also contribute to understanding of other inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of sarcoidosis
* Swedish speaking
* Able to understand and approve of study protocol
* No contraindications for planned interventions

Exclusion Criteria:

* No suspicion of sarcoidosis
* Not Swedish-speking
* Not able to understand study protocol
* Not approving of stydy protocol
* Contraindications for planned interventions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2034-05-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
Immune cell percentages in lung, lymph nodes and blood | 2 years
  Is there a difference in frequency of different immune cells (percentage) between different compartments in clinical disease phenotypes?

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden